CLINICAL TRIAL: NCT07255326
Title: Role of Omega-3 Fatty Acids in Modulating Retinal Microvascular Changes in Type 1 Diabetes
Brief Title: Effect of Omega-3 Fatty Acids on Eye Blood Vessels in Type 1 Diabetes
Acronym: O3RETINA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Faisalabad (Other)
Responsible Party: Principal Investigator, Nida Amin, Assistant Professor/HOD Optometry Department, University of Faisalabad
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NIDA_OMEGA3_T1D_RETINA_001; 1174/CH-UCHS (Other: The Children's Hospital & University of Child Health Sciences, Lahore)
Record Dates: First submitted 2025-11-14; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Diabetic Retinopathy; Type 1 Diabetes; Omega 3 Fatty Acids
Keywords: Diabetic retinopathy; retinal microvasculature; omega 3 fatty acids; type 1 diabetes
MeSH Terms: conditions — Diabetic Retinopathy; Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either the omega-3 supplement group or a control group that does not receive the supplement. Both groups will attend regular eye exams every three months to monitor changes in retinal blood vessels. Outcomes will be compared between the two groups to assess the effects of omega-3 supplementation
Who Masked: Participant, Care Provider, Investigator
Masking Description: Laboratory staff analyzing blood samples and retinal imaging technicians will be blinded to group assignments
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omega-3 Supplement Group (Experimental): Participants will take one daily capsule containing 1000 mg of combined EPA and DHA. The supplement is taken orally with food. Eye exams will be performed every three months to monitor retinal blood vessel health.
  Interventions: Dietary Supplement: Omega 3 Fish Oil supplements
- Omega-3 Control Group (Placebo Comparator): Participants will take a daily capsule that looks identical to the omega-3 supplement but contains no active omega-3 fatty acids. Eye exams will be performed every three months to monitor retinal blood vessel health. Participants will report any health changes.
  Interventions: Dietary Supplement: Omega 3 Fish Oil supplements

INTERVENTIONS:
Dietary Supplement: Omega 3 Fish Oil supplements — Arm 1 - Omega-3 Supplement Group:
  Intervention Type: Dietary Supplement Intervention Name: Omega-3 Fatty Acid Supplement
  Intervention Description:
  Participants will take one daily capsule containing 1000 mg of combined EPA and DHA. The supplement is taken orally with food. Eye exams will be performed every three months to monitor retinal blood vessel health. Participants will report any side effects such as mild stomach upset.
  Arm 2 - Placebo / Control Group:
  Intervention Type: Placebo Intervention Name: Placebo Capsule
  Intervention Description:
  Participants will take a daily capsule that looks identical to the omega-3 supplement but contains no active omega-3 fatty acids. Eye exams will be performed every three months to monitor retinal blood vessel health. Participants will report any health changes.
  Other Names: Placebo

SUMMARY:
The aim of this clinical trial is to learn if omega-3 fatty acid supplements help maintain healthy blood vessels in the eyes of adults with type 1 diabetes. It will also learn about the safety of omega-3 supplements. The main questions it aims to answer are:

Do omega-3 supplements improve the health of retinal blood vessels in adults with type 1 diabetes? Are there any side effects when taking omega-3 supplements? Researchers will compare participants taking omega-3 supplements to a control group (if applicable) to see if the supplements help support retinal blood vessel health.

Participants will:

Take a daily omega-3 supplement for the duration of the study Attend regular eye exams to monitor changes in the retina Report any side effects or health changes during the study

DETAILED DESCRIPTION:
People with type 1 diabetes are at risk of having changes in microvasculature of the retina, which may impair visual functions with time. This paper examines the potential of daily supplemental intake of omega -3 fatty acids to maintain retinal vascularity and prevent the ocular complications linked to diabetes. The researchers seek to know whether the supplements can protect the eyes and enhance the long-term eye health.

The trial participants will consume a daily dose of omega 3 and visit a clinic after every quarterly interval to take ophthalmic tests. In the process of such appointments the research team will examine the health of the retinal and record any vascular changes. Another questionnaire that will be administered to the participants is the one that focuses on adverse events, including mild gastrointestinal discomfort, linked to supplementation.

The trial period will take around 12 months. The control cohort will be assigned to the non-supplemented group in order to compare the differences in retinal microvascular health in subjects subjected to omega-3 supplementation. The results although may not have immediate therapeutic value would inform future interventions to prevent or mitigate ocular complications in people with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of Type 1 Diabetes Age between 10 and 45 years Duration of diabetes ≥ 2 years Mild to moderate diabetic retinopathy allowed (based on fundus examination)

Exclusion Criteria:

Presence of any ocular disease other than diabetic retinopathy Use of medications that may affect retinal vascular measurements or visual function outcomes Presence of systemic diseases other than diabetes (e.g., uncontrolled hypertension, autoimmune diseases) History of ocular surgery within the past 6 months Current participation in another interventional clinical trial

Ages: 10 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Change in Retinal Artery Diameter | 3 Months
  Change in central retinal artery equivalent measured from fundus photographs using OCTA
Change in Retinal Vein Diameter | 3 Month
  Change in central retinal vein equivalent measured from fundus photographs using OCTA
Change in Arterio-Venous Ratio | 3 months
  Change in AVR calculated automatically as CRAE divided by CRVE

SECONDARY OUTCOMES:
Change in Best-Corrected Visual Acuity | 3 Months
  Change in BCVA measured using the logMAR chart at 4 meters
Change in Contrast Sensitivity | 3 Months
  Change in contrast sensitivity measured using the Pelli-Robson chart
Change in HbA1c | 3 Months
  Change in glycosylated hemoglobin (HbA1c) measured through laboratory blood testing
Change in Fasting Blood Glucose | 3 Months
  Change in fasting blood glucose measured through venous blood sampling

CONTACTS AND LOCATIONS:
Locations (1):
- Children Hospital Lahore and Ali Fatima Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data will not be shared publicly. Summary-level results will be published in peer-reviewed journals and may be shared with researchers upon reasonable request. Study protocol, statistical analysis plan, and informed consent form may be available upon request from the principal investigator. Researchers can contact the principal investigator for data access requests.

REFERENCES:
- [Result] Sala-Vila A, Vinagre I, Cofan M, Lazaro I, Ale-Chilet A, Barraso M, Hernandez T, Harris WS, Zarranz-Ventura J, Ortega E. Blood omega-3 biomarkers, diabetic retinopathy and retinal vessel status in patients with type 1 diabetes. Eye (Lond). 2025 Jun;39(8):1526-1531. doi: 10.1038/s41433-025-03705-5. Epub 2025 Feb 18. PMID 39966603
- [Result] Elbarbary NS, Ismail EAR, Mohamed SA. Omega-3 fatty acids supplementation improves early-stage diabetic nephropathy and subclinical atherosclerosis in pediatric patients with type 1 diabetes: A randomized controlled trial. Clin Nutr. 2023 Dec;42(12):2372-2380. doi: 10.1016/j.clnu.2023.10.007. Epub 2023 Oct 13. PMID 37862823
- See also: Official research portal of The University of Faisalabad, the sponsoring institution for this PhD study. — https://tuf.edu.pk/
- See also: The Children's Hospital & Institute of Child Health, Lahore — https://chich.edu.pk/